CLINICAL TRIAL: NCT06617975
Title: Evaluation of the Effectiveness of the Spa Therapy Program for Rheumatology at Santenay in Patients With Knee Osteoarthritis
Brief Title: Knee Osteoarthritis and Spa Therapy
Acronym: SANTIAGO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CEN Biotech (Industry)
Collaborators: COMPAGNIE EUROPEENNE DES BAINS (Unknown); VALVITAL Santenay (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: C1729
Record Dates: First submitted 2024-09-23; First posted 2024-10-01 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Knee Osteoarthritis; Knee Osteoarthritis (OA)
Keywords: Balneotherapy; Spa therapy; Rheumatology; Knee osteoarthritis; WOMAC
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Prospective, single-arm, superiority study with external comparison (control group of a reference RCT)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Balneotherapy (Experimental): 18-day balneotherapy program with Mineral Water of Santenay in addition to standard of care for knee osteoarthritis
  Interventions: Other: Balneotherapy program in rheumatology indication

INTERVENTIONS:
Other: Balneotherapy program in rheumatology indication — At least 4 balneotherapy sessions per day, 6 days a week during 3 consecutive weeks that may include: 1 whirlpool bath per day, 1 poultice application per day, 1 bath with immersion showers in a pool per day, a local jet shower every other day, a penetrating shower every other day.
  Alternative treatments may replace penetrating shower or local jet shower, or other care, e.g., collective jet shower or steam bath. 10-minute air diffusion baths are taken in individual tubs at 37°C. Mud is applied 10 minutes as a poultice to both knees (minimum 2 per knee, 52°C), if necessary, to other painful osteoarthritis areas. 10-minute collective pool bathing takes place in a thermal pool equipped with jet stations immersed in water at 32°C. 3-minute local jet shower is applied to the predefined area using thermal water at 37°C. 10-minute penetrating showers are delivered by an affusion ramp on the patient lying down and directed on the area defined, using thermal water at 37°C.

SUMMARY:
The aim of this clinical trial is to assess the efficacy of the 18-day balneotherapy program (therapeutic indication: Rheumatology) in terms of functional incapacity and the disorders (pain, joint stiffness) induced by osteoarthritis of the knee, and thus improves patients' quality of life, in patients presented with knee osteoarthritis.

The French National Academy of Medicine encourages the re-use of RCT data when available. In this context, the current study is designed as a single-arm prospective study with external comparison using the propensity score. The Control group consists of the patients which were allocated to the Control group of reference randomized clinical trial (RCT) "ANGELLO Study" (NCT05819437). These patients received standard care for knee osteoarthritis, i.e., pain management and exercise recommendations.

All patients enrolled in the current study benefit of 18-day balneotherapy program (therapeutic indication: Rheumatology) with Mineral Water of Santenay (Burgundy, France), and examination with a practitioner at enrollment and 6 months after the beginning of spa treatment.

DETAILED DESCRIPTION:
For study purposes, two medical visits with the investigator are organized: the first in the 28 days preceding the 18-day balneotherapy program, or at the latest on the first day of the program, before the first care, and the second 6 months after the start of the program. A remote visit at 3 months is also organized.

The data required for study evaluations are collected by the investigator or self-evaluated by patients during the visits.

Patients of the study receive the same exercise recommendations than the patients of the Control group of the reference study, and their body weight as well as physical ability are monitored.

ELIGIBILITY:
Inclusion Criteria:

* Knee osteoarthritis with Kellgren and Lawrence stage 2 to 4 evidenced by a knee X-ray examination in the past 3 years.
* 100-normalized score of the WOMAC physical function subscale greater than or equal to 30.
* Accepting a prescription for a balneotherapy program in the Rheumatology at Santenay spa as part of the management of their knee osteoarthritis issued by the investigator.
* Signed inform consent.
* With health insurance affiliation.

Exclusion Criteria:

* Presented with balneotherapy contraindication or to certain adjuvant treatment techniques (balneation, hydrotherapy jets, massage): chronic infectious pathology, active cancer, decompensated cardiac, hepatic or renal insufficiency, "open" leg ulcer, immune deficiency, phlebitis, erysipelas or history of erysipelas, active thrombosis, behavioral disorders, etc.
* Presented with chronic pain for reasons other than osteoarthritis: chronic inflammatory rheumatism (rheumatoid arthritis, ankylosing spondylitis, lupus, psoriatic arthritis) or fibromyalgia.
* Having had spa treatment in the past 6 months whatever the indication or intra-articular corticosteroid injection within the previous 90 days or hyaluronic acid infiltration within the previous 6 months.
* Having planned a spa treatment in another indication between inclusion and final visit.
* Patient scheduled for knee osteoarthrosis-related surgery within the next 7 months.
* Residing more than 30 kilometers from Santenay at the time of spa treatment. Women of childbearing potential who are not using effective contraception (estrogen/progestin or progestin-only oral, vaginal, transdermal, injectable or subcutaneous) or who plan to discontinue contraception within the next 7 months.
* Likely to be unable to comply with protocol or to attend visits, particularly in view of the duration of the research, or unable to read or understand French.
* Regulatory reason (guardianship or already enrolled in a clinical trial).
* Already included in a clinical trial or in the exclusion period of a clinical trial.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-10-14 (Actual); Primary Completion 2026-12-15 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Minimal Clinically Important Improvement (MCII) at 6 months | 6 months
  MCII is defined as a pain reduction of 19.9 mm or more on a 0-100 visual analogic scale (VAS), where 0 means no pain and 100 worse pain.
  The percentage of patients achieving MCII is calculated and compared with that of the control group in the reference RCT (external comparison).
Minimal Clinically Important Improvement (MCII) at 6 months | 6 months
  MCII is defined as a reduction of 9.1 points or more in the function subscale of the Physical function subscale of the Western Ontario and McMaster Universities Arthritis Index (WOMAC) in absence of knee surgery. WOMAC is a self-administered questionnaire that consists in 17 items: (17 items): using stairs, rising from sitting, standing, bending, walking, getting in / out of a car, shopping, putting on / taking off socks, rising from bed, lying in bed, getting in / out of bath, sitting, getting on / off toilet, heavy domestic duties, light domestic duties. The 100-normalized subscale score ranges from 0 (none) to 100 (worse functional limitations).
  The percentage of patients achieving MCII is calculated and compared with that of the control group in the reference RCT (external comparison).

SECONDARY OUTCOMES:
Change from baseline of pain-related knee osteoarthritis at 3 months | Day 1 and 3 months
  Pain intensity is measured using a 0 (no pain)-100 (Worse pain) Visual Analogic Scale (VAS). Mean variation is compared with that of the control group in the reference RCT (external comparison).
Change from baseline of pain-related knee osteoarthritis at 6 months | Day 1 and 6 months
  Pain intensity is measured using a 0 (no pain)-100 (Worse pain) Visual Analogic Scale (VAS). Mean variation is compared with that of the control group in the reference RCT (external comparison).
Change from baseline of the pain subscale of the WOMAC at 3 months | Day 1 and 3 months
  Pain subscale of the WOMAC is a self-administered questionnaire that consists in 5 items: during walking, using stairs, in bed, sitting or lying, and standing upright. The 100-normalized subscale score ranges from 0 (none) to 100 (worse pain limitations). Mean variation is compared with that of the control group in the reference RCT (external comparison).
Change from baseline of the pain subscale of the WOMAC at 6 months | Day 1 and 6 months
  Pain subscale of the WOMAC is a self-administered questionnaire that consists in 5 items: during walking, using stairs, in bed, sitting or lying, and standing upright. The 100-normalized subscale score ranges from 0 (none) to 100 (worse pain limitations). Mean variation is compared with that of the control group in the reference RCT (external comparison).
Changes from baseline of stiffness subscale of the WOMAC at 3 months | Day 1 and 3 months
  Stiffness subscale of the WOMAC is a self-administered questionnaire that consists in 2 items: during walking, using stairs, in bed, sitting or lying, and standing upright. The 100-normalized subscale score ranges from 0 (none) to 100 (worse stiffness limitations). Mean variation is compared with that of the control group in the reference RCT (external comparison).
Changes from baseline of stiffness subscale of the WOMAC at 6 months | Day 1 and 6 months
  Stiffness subscale of the WOMAC is a self-administered questionnaire that consists in 2 items: during walking, using stairs, in bed, sitting or lying, and standing upright. The 100-normalized subscale score ranges from 0 (none) to 100 (worse stiffness limitations). Mean variation is compared with that of the control group in the reference RCT (external comparison).
Change from baseline of physical function subscale of the WOMAC at 3 months | Day 1 and 3 months
  Physical function subscale of the Western Ontario and McMaster Universities Arthritis Index (WOMAC) is a self-administered questionnaire that consists in 17 items: (17 items): using stairs, rising from sitting, standing, bending, walking, getting in / out of a car, shopping, putting on / taking off socks, rising from bed, lying in bed, getting in / out of bath, sitting, getting on / off toilet, heavy domestic duties, light domestic duties. The 100-normalized subscale score ranges from 0 (none) to 100 (worse functional limitations). Mean variation is compared with that of the control group in the reference RCT (external comparison).
Change from baseline of physical function subscale of the WOMAC at 6 months | Day 1 and 6 months
  Physical function subscale of the Western Ontario and McMaster Universities Arthritis Index (WOMAC) is a self-administered questionnaire that consists in 17 items: (17 items): using stairs, rising from sitting, standing, bending, walking, getting in / out of a car, shopping, putting on / taking off socks, rising from bed, lying in bed, getting in / out of bath, sitting, getting on / off toilet, heavy domestic duties, light domestic duties. The 100-normalized subscale score ranges from 0 (none) to 100 (worse functional limitations). Mean variation is compared with that of the control group in the reference RCT (external comparison).
Change from baseline of total score of the WOMAC at 3 months | Day 1 and 3 months
  The scores for each of the 3 subscales (function, pain, stiffness) are summed up to calculate the total WOMAC score. The 100-normalized score ranges from 0 (none) to 100 (worse limitations).
Change from baseline of total score of the WOMAC at 6 months | Day 1 and 6 months
  The scores for each of the 3 subscales (function, pain, stiffness) are summed up to calculate the total WOMAC score. The 100-normalized score ranges from 0 (none) to 100 (worse limitations).
Acceptable Symptom State (ASS) at 3 months | 3 months
  ASS is defined as VAS pain value of 32 mm or less or a WOMAC function subscale, normalized to a 0-100 score of 31 points or less. The percentage of patients achieving ASS is calculated and compared with that of the control group in the reference RCT (external comparison).
Acceptable Symptom State (ASS) at 6 months | 6 months
  ASS is defined as VAS pain value of 32 mm or less or a WOMAC function subscale, normalized to a 0-100 score of 31 points or less. The percentage of patients achieving ASS is calculated and compared with that of the control group in the reference RCT (external comparison).
Changes from baseline of quality of life at 3 months | Day 1 and 3 months
  Quality of life is measured using EUROQOL (EQ-5D-3L) questionnaire. The EQ-5D-3L descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results into a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes patient health state. Mean variation is compared with that of the control group in the reference RCT (external comparison).
Changes from baseline of quality of life at 6 months | Day 1 and 6 months
  Quality of life is measured using EUROQOL (EQ-5D-3L) questionnaire. The EQ-5D-3L descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results into a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient health state. Mean variation is compared with that of the control group in the reference RCT (external comparison).
Management of knee osteoarthritis over the study | 6 months
  Number and frequency of treatments for knee osteoarthritis (analgesics, chondro-protectors or antarthritics, intra-articular injections of corticoids and hyaluronic acid, physical or surgical treatments). Numbers and frequencies of treatments are compared with those of the control group in the reference RCT (external comparison).
Safety of the18-day balneotherapy program (therapeutic indication: Rheumatology) at Santenay | 6 months
  Adverse effects related to the 18-day balneotherapy program (therapeutic indication: Rheumatology) with Santenay mineral water are described using MedDRA, whether they occurred during or after the program.

OTHER OUTCOMES:
Satisfaction with the spa therapy and spa site | Day 18
  Subjective opinion of patients regarding spa cares, facilities and staff, is collected at the end of the program, and measured using a 5-point Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno COLLOMBIER, MD, Principal Investigator
Locations (1):
- Valvital - Thermes de Santenay, Santenay, Burgundy, France

IPD SHARING:
Plan to Share IPD: Undecided
Patient data is not anonymized. To comply with European regulations and national provisions, patients are informed that no sharing of IPD is planned in order to protect their personal data. If data is to be shared, patients must be informed individually and their consent obtained.
  At this stage, only aggregated data can be shared.

REFERENCES:
- See also: ANGELLO STUDY — https://clinicaltrials.gov/study/NCT05819437